CLINICAL TRIAL: NCT04665726
Title: Natural History Study of Usher Syndrome in a Cohort of Patients Followed Longitudinally for 5 Years
Brief Title: Natural History Study of Usher Syndrome ( Light4Deaf )
Acronym: Light4Deaf
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P16-05; 2016-A01715-46 (Other: N°IDRCB)
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Usher Syndromes
Keywords: Usher syndrome,; Natural history study for retinal degenetation,; Deep-phenotyping,; Hearing loss,; Vestibular dysfunction
MeSH Terms: conditions — Usher Syndromes; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA, skin fibroblasts for future disease modelling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical centres in the LIGHT4DEAF consortium have developed and will continue to improve a reliable, early molecular diagnosis and protocols for full clinical characterisation of Usher syndrome, which will be valuable for the foreseen USH clinical trials. The clinical arm of the project aims at performing a deep-phenotyping of retinal degeneration, hearing loss, vestibular dysfunction, neurocognitive ability of subects with a molecular diagnosis of any Usher syndrome. Functional and structural parameters for retinal, auditory, and vestibular impairments are followed overtime to document the natural history of the disease and establish relevant clinical endpoint for disease progression that may be useful for future clinical trials.

DETAILED DESCRIPTION:
Our cohort study aims at precisely documenting ophthalmic, auditory, vestibular, cogninitive alterations over time with phenotype/genotype correlation Ophthalmological assessment; Best corrected visual acuity, kynetic perimetry, microperimetry, colour contrast sensitivity, retinal multimodal imaging (fundus photograph, fundus autofluorescence, SD-OCT, OCTA, adaptive optics)

ENT assessment:

Tone and voice audiometry, Distortion product otoacoustic emissions Language assessment for children

Vestibular assessment:

Complete assessment of vestibular, canal and otolithic function Neuro-cognitive and visio spatial assessment Genetic: deep-genotyping using next generation sequencing

ELIGIBILITY:
Inclusion Criteria:

* Patient with a molecular diagnosis of Usher syndrome type I, II or III or a clinical diagnosis of Usher syndrome type I, II or III which will then be confirmed by a molecular diagnosis
* Health insurance beneficiary
* Informed consent signed by the patient or their legal representatives

Exclusion Criteria:

• Patient or his/her legal representatives unable to understand the study and for whom informed consent cannot be obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient affected with Usher syndrome that has been molecularly confirmed
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2022-06-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
5-year natural history of Usher syndrome | From date of inclusion until the date of last documented progression , assessed up to 5 years
  Phenotype/genotype correlation, structure function correlation and progression of structural and functional parameters

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AUDO, Pr, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (4):
- France (4):
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - CHU Pitié Salpêtrière, Paris
  - CHU Necker, Paris
  - CHU Robert Debré, Paris